CLINICAL TRIAL: NCT01994395
Title: Randomized Control Trial Comparing Walking Task Specific Training With Stride Management Assist (SMA) Device vs.Functional Task Specific Training on Functional Walking Ability in Outpatient Stroke Rehabilitation
Brief Title: Development of Walk Assist Device to Improve Community Ambulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Honda (Unknown)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUSTU00085161
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: Stroke; Gait; Stride Management Assist; Mild-moderate Stroke, post 30 days or longer
MeSH Terms: conditions — Stroke | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The SMA group (task specific training) will be trained to simulate the demands of overground walking. The impairment based group will match the SMA group in intensity but will be focused on balance and other functional goals rather than explicitly on walking. The rationale of this study is to assess task specific training with SMA vs. impairment based training. To this end, we will use the Stride Management Assist device by Honda Corporation and compare it to impairment based physical therapy in outpatient sessions.
Who Masked: Outcomes Assessor
Masking Description: A blinded research physical therapist will test the outcome measure at baseline, Mid Testing after Session 9 , at Post Testing after Session 18 and at 3 month follow up testing after Session 18.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stride Management Assist (SMA) System (Experimental): Participants will be randomized into either the SMA group or impairment based (IPT) group. The SMA group (task specific training) will be trained to simulate the demands of overground walking using the Stride Management Assist Device in outpatient physical therapy.
  Interventions: Device: The Stride Management Assist (SMA) System
- Impairment based therapy (Active Comparator): Impairment based therapy will include traditional functional mobility training physical therapy. It will match the SMA group in intensity but will be focused on balance and other functional goals rather than explicitly on walking in outpatient physical therapy.
  Interventions: Other: Impairment based therapy

INTERVENTIONS:
Device: The Stride Management Assist (SMA) System — Participants will participate in 18 sessions of outpatient physical therapy + 3 sessions of testing for up to 8 weeks. Assessment (strength, flexibility, balance, sensation, endurance, transfers, gait. Treatment consists of 30 minutes high intensity gait training with device, 15 minutes functional mobility with device.
  Arms: Stride Management Assist (SMA) System
Other: Impairment based therapy — Participants participate in 18 weeks of outpatient physical therapy + 3 assessment sessions. Assessment (strength, flexibility, balance, sensation, endurance, transfers, gait). Treatment will be divided into: 15 min balance training, 15 minutes functional mobility (transfers, strength or flexibility training) and 15 min high intensity gait training
  Arms: Impairment based therapy

SUMMARY:
Hypothesis/Specific Aims:

The purpose of this study is to determine the effect of training with the Stride Management Assist (SMA) device vs. Impairment based physical therapy (IPT) on descending corticospinal drive to the lower limb muscles in patients post stroke. The investigators hypothesize that long-term SMA use would strengthen the connections between the motor areas of the brain and the lower limbs. Specifically, individuals in the SMA group will show higher corticospinal excitability of the lower limb muscles compared to those in the IPT group.

DETAILED DESCRIPTION:
This is a randomized control trial comparing task specific training with the Stride Management Assist (SMA) device verses an impairment based physical therapy (IPT) approach on functional walking ability in outpatient stroke rehabilitation. Participants between the ages of 18-80 and who are 30 days or greater post stroke will be included.

This SMA robotic device assists hip flexion and extension, for each side independently. It is controlled through software run on a tablet. The device weighs 2.8 kgs, and has 2 brushless direct current motors running on a rechargeable lithium ion battery. It comes in 3 sizes (small, medium and large). It is worn around like a belt with the motors near the hips and straps on the thighs. The SMA device allows users to increase their stride length by providing assist with the motors in flexion and extension. This device is 1) simple to use in the clinical setting; 2) easily adjustable to alter according to the requirements of each subject; and, 3) can quantify the amount of assistance required to facilitate walking patterns.

Participants post stroke 30 days or greater will be recruited from inpatient, day rehabilitation and outpatient clinics. Participants will be scheduled for 18 Sessions of outpatient physical therapy plus 3 sessions of testing. The amount of sessions provided will be dependent upon compatibility with the device and ability to tolerate the device. A participant will continue with each session of the study as deemed appropriate by research staff.

* A. Phase I. (session 0): After consenting, subjects will undergo a physical evaluation and screening exam by a licensed physical therapist. If they meet study criteria, they will be randomly placed into either the SMA group or the IPT group using a random number generator and they will be entered into the study. Once they are enrolled, baseline outcome measures will be assessed by a blinded research physical therapist.
* B. Phase II. (sessions 1-9):

  * Stride Management Assist Group: Treatment consists of 30 minutes high intensity gait training with device, 15 minutes functional mobility with device.
  * Impairment Based Physical Therapy Group: Treatment will be divided into: 15 min balance training, 15 minutes functional mobility (transfers, strength or flexibility training) and 15 min high intensity gait training
* C. Phase III. (session 10): Mid treatment assessment. Outcome measures will be assessed by a blinded research physical therapist.
* D. Phase II. (sessions 11-19):

  * Stride Management Assist Group: Treatment consists of 30 minutes high intensity gait training with device, 15 minutes functional mobility with device.
  * Impairment Based Physical Therapy Group: Treatment will be divided into: 15 min balance training, 15 minutes functional mobility (transfers, strength or flexibility training) and 15 min high intensity gait training
* E. Phase IV. (session 20): Post Testing. Outcome measures will be assessed by a blinded research physical therapist.

All testing and training sessions will be under the supervision of a licensed physical therapist. All subjects will be permitted to stop physical activity or rest at any time during the study. Adverse events will be recorded.

The investigators anticipate this study will help determine if the Stride Management Assist is a practical option to better strengthen the connections between the brain and the lower limbs. The investigators do not foresee any potential pitfalls.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30-days post stroke
* Initial gait speed of > 0.4 m/s and < 0.8 m/s
* Adequate cognitive function (MMSE score >17)
* Subject is willing to be randomized to the control group or the treatment group.
* Ability to sit unsupported for 30 seconds
* Ability to walk at least 10m with maximum 1 person assist,
* Ability to follow a three-step command
* Physician approval for patient participation
* Living in the community post-stroke with ability to travel to the intervention site to participate in the outpatient program and able to perform the home exercise program in the residential facility.
* Willing to carry wireless body sensors through the period of the study and to follow-up time period, post inpatient stroke, cardiac, pulmonary, or any other lower extremity physical rehabilitation
* ≥ 90 days post major orthopedic surgery (i.e. hip, knee, and/or ankle joint replacement)
* ≥ 6 months post coronary artery bypass grafting (CABG) or cardiac valve procedure
* Able and willing to give written consent and comply with study procedures, including follow-up visits
* Cannot not be participating in any other structured outpatient or home health physical therapy program

Exclusion Criteria:

* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* Severe arthritis or orthopedic problems that limit passive ranges of motion (ROM) of lower extremity (knee flexion contracture of > 10°, knee flexion ROM < 90°, hip flexion contracture > 25°, and ankle plantar flexion contracture > 15
* Serious medical conditions including myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living, Severe hypertension, severe weight bearing pain, life expectancy less than one year
* Preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia
* History of major head trauma, Lower extremity amputation, Non-healing ulcers of a lower extremity, Renal dialysis or end stage liver disease, Legal blindness or severe visual impairment, a history of significant psychiatric illness
* History of unexplained, recurring headaches, epilepsy/seizures/skull fractures or skull deficits
* Medications that lower seizure threshold
* History of concussion in last 6 months
* Subject is pregnant, nursing or planning a pregnancy
* Inability to travel 3 times per week for outpatient training programs
* Participating in another clinical trial that, according to the Principal Investigator, is likely to affect study outcome or confound results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayaraman A, O'Brien MK, Madhavan S, Mummidisetty CK, Roth HR, Hohl K, Tapp A, Brennan K, Kocherginsky M, Williams KJ, Takahashi H, Rymer WZ. Stride management assist exoskeleton vs functional gait training in stroke: A randomized trial. Neurology. 2019 Jan 15;92(3):e263-e273. doi: 10.1212/WNL.0000000000006782. Epub 2018 Dec 19. PMID 30568009
- [Derived] Buesing C, Fisch G, O'Donnell M, Shahidi I, Thomas L, Mummidisetty CK, Williams KJ, Takahashi H, Rymer WZ, Jayaraman A. Effects of a wearable exoskeleton stride management assist system (SMA(R)) on spatiotemporal gait characteristics in individuals after stroke: a randomized controlled trial. J Neuroeng Rehabil. 2015 Aug 20;12:69. doi: 10.1186/s12984-015-0062-0. PMID 26289955

RESULTS

PARTICIPANT FLOW:
Groups:
- Stride Management Assist (SMA) System: Participants will be randomized into either the SMA group or impairment based (IPT) group.
  The Stride Management Assist (SMA) System: Participants will participate in 18 sessions of outpatient physical therapy + 3 sessions of testing for up to 8 weeks. Assessment (strength, flexibility, balance, sensation, endurance, transfers, gait. Treatment consists of 30 minutes high intensity gait training with device, 15 minutes functional mobility with device.
- Impairment Based Therapy: Impairment based therapy will include traditional functional mobility training physical therapy.
  Impairment based therapy: Participants participate in 18 weeks of outpatient physical therapy + 3 assessment sessions. Assessment (strength, flexibility, balance, sensation, endurance, transfers, gait). Treatment will be divided into: 15 min balance training, 15 minutes functional mobility (transfers, strength or flexibility training) and 15 min high intensity gait training
Period: Overall Study
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Started | 26 | 27
Completed | 25 | 25
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: One subject dropped out at baseline screening, prior to assignment to any group. One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 6 | 11 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
  years
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 60 (10) | 62 (13) | 61 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
  Participants
    number analyzed (Participants) | 25 | 25 | 50
    Female | 8 | 9 | 17
    Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
  participants
    United States: number analyzed (Participants) | 25 | 25 | 50
    United States | 25 | 25 | 50
10 Meter Walk Test [Mean (Standard Deviation); unit: meters per second] — Study criteria require initial gait speed of > 0.4 m/s and < 0.8 m/s Participants were asked to walk at their normal self-selected speed 14 meters and the time is measured for the intermediate 10 meters to allow for acceleration and deceleration. This is repeated for three trials and then averaged. Population: One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
  meters per second
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 0.7 (0.1) | 0.65 (0.1) | 0.68 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in 10 Meter Walk Test From Baseline in Gait Speed
Description: Measure of self selected and fast walking speeds by measuring the time it takes an individual to walk 10 meters. The test is performed using a "flying start," patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go." and repeated "Please walk this distance as fast as you can safely when I say go."
Time Frame: Baseline Assessment (Visit 1), Mid Training Assessment (Visit 10), Post Training Assessment (Visit 18), 3 Month Post Training Assessment (3 Month Follow-up)
Population: One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
meters per second
  Baseline Assessment | 0.7051 (0.122677) | 0.6606 (0.12067815)
  Mid Training Assessment | 0.8544 (0.202805061) | 0.7547 (0.16119851)
  Post Training Assessment | 0.9566 (0.20176847) | 0.8376 (0.191048354)
  3 Month Post Training Assessment | 0.9439 (0.226535699) | 0.8085 (0.169381067)

2. Secondary Outcome: Activities-Specific Balance Confidence Scale (ABC)
Description: ABC is a 16-item self-report measure in which patients rate their balance confidence in performing various ambulatory activities without falling. Items are rated on a scale ranging from 0-100, with zero representing no confidence and 100 representing complete confidence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 66.7625 (18.00944) | 67.6472 (17.7136527)
  Mid Training Assessment | 73.2067 (15.44828) | 70.4443 (17.4234304)
  Post Training Assessment | 79.1630 (13.30643987) | 77.99 (13.3571932)
  3 Month Post Training Assessment | 81.6292 (11.41238) | 78.3749 (13.50986798)

3. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: The NPRS is an 11-point scale from 0-10 where patients verbally select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours from 0 (no pain) to 10 (the most intense pain imaginable).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 0.733336 (1.589901) | 0.680004 (1.67631206)
  Mid Training Assessment | 1.166668 (1.83081) | 0.72458 (1.61792765)
  Post Training Assessment | 0.879996 (1.83081) | 0.599995 (1.45295656)
  3 Month Post Training Assessment | 1.568606 (2.136855) | 0.587721053 (1.235250407)

4. Secondary Outcome: Stroke Specific Quality of Life Scale (SS-QOL)
Description: A 49 item assessment grouped into 12 domains of health-related quality of life in stroke survivors; including areas of mobility, energy, upper extremity function, work and productivity, mood, self-care, social roles, family roles, vision, language, thinking, personality. Each individual domain consists of 3 to 10 items that are averaged to generate an overall score, each item is rated on a 5- point Likert scale, with a minimum value of 1 (meaning the worst outcome) and a maximum value of 5 (meaning the best outcome). Domains scores (non-weighted average of item scores) and a summary score (non-weighted average of all 12 domain scores) are computed. Summary scores range from 49-245, with higher scores indicating better functioning.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 198.16 (21.30665) | 193.84 (25.4945746)
  Mid Training Assessment | 204.8 (23.02897) | 205.36 (23.5741384)
  Post Training Assessment | 205.6 (24.54248018) | 211.72 (23.3158029)
  3 Month Post Training Assessment | 200.3529 (25.22633) | 211.5789474 (27.31771055)

5. Secondary Outcome: The Modified Falls Efficacy Scale (mFES)
Description: 14 item questionnaire assessing individuals' confidence in their ability to perform tasks without falling. Individuals rate their confidence from 0 (not confident at all) to 100 (completely confident).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 8.3803 (1.448756) | 8.4426 (1.20545002)
  Mid Training Assessment | 8.9228 (1.061062) | 8.719996 (0.98649669)
  Post Training Assessment | 9.0971 (0.937882386) | 9.075176 (0.9848385)
  3 Month Post Training Assessment | 9.2941 (0.785258) | 9.078111111 (1.094633589)

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: PHQ-9 is a 9-item self-report questionnaire designed to diagnose both the presence of depressive symptoms as well as to characterize the severity of depression. A single question rates how difficult problems have made it to do work, take care of things at home or get along with other people using a 4 level scale (not difficult at all to extremely difficult). Each item is scored from 0-3; total scores may be 0-27, with higher scores representing increased severity of depression.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 3.72 (3.553402) | 3.68 (4.31779265)
  Mid Training Assessment | 2.88 (2.437895) | 3.12 (4.12633817)
  Post Training Assessment | 2.32 (2.267891826) | 2.16 (3.15805848)
  3 Month Post Training Assessment | 3.352941 (2.935583) | 2.631578947 (2.8908000088)

7. Secondary Outcome: Participants Receiving Transcranial Magnetic Stimulation (TMS)
Description: To compare the effect of training on the connections between the brain and leg muscles (descending corticomotor drive) using a non-invasive brain stimulation called transcranial magnetic stimulation (TMS). TMS is a safe, non-invasive, painless method of brain stimulation that has been widely used to study the physiology of the representations of muscles in the motor cortex in healthy and neurologically disordered individuals13. Very short duration (< 1 ms) magnetic pulses are applied via an insulated wire coil placed on the intact scalp overlaying the motor cortical area projecting to a target muscle. Each pulse induces a motor evoked potential (MEP) in a target muscle that can be readily monitored by recording Electromyogram (EMG) from that muscle. A figure-of-eight or double cone coil is typically used to deliver focal magnetic pulses to a number of scalp sites over the cortical area representing a muscle of interest.
Time Frame: Session 0 (initial visit);Session 20 (between 6-8 weeks)
Population: One subject dropped before being assigned to a group. One subject from SMA group and 2 from impairment based therapy group dropped due to scheduling conflicts prior to starting any training.
Measure: Count of Participants; unit: Participants
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
Participants
  Session 0 | 15 | 15
  Session 20 | 15 | 15

8. Secondary Outcome: Change in 6 Minute Walk Test From Baseline in Distance (6MWT)
Description: The 6 Minute Walk Test (6MWT) is a test of endurance, by measuring the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary.The distance is measured with a measuring wheel. The instructions are "Walk covering as much ground as you can in 6 min. You can stop to sit or stand if needed, but time will keep running." The change in the distance walked in the 6-minute walk can be used to evaluate the efficacy of an exercise-training program or to trace the natural history of change in exercise capacity over time. The 6MWT is measured in meters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre Training Assessment | 874.6067 (220.4362) | 794.33 (151.703575)
  Mid Treatment Assessment | 1140.5040 (364.1122684) | 963.1633 (227.048913)
  Post Training Assessment | 1268.24 (344.0931699) | 1065.5567 (227.1440369)
  3 Month Post Training Assessment | 1230.3088 (375.9471237) | 1035.1053 (185.5663909)

9. Secondary Outcome: Berg Balance Scale (BBS)
Description: The BBS is a 14-item objective measure designed to assess static balance and fall risk in adult populations and is a well-accepted measure in the stroke literature. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed. Each item is scored from 0 to 4 points. The maximum score is 56 points. A score from 0 to 20 represents balance impairment, 21 to 40 represents acceptable balance, and 41-56 represents good balance. The minimal detectable change score for individuals with acute stroke is 6.9 points16 and 4.66 points in chronic stroke17.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale, each item scored 0-4
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
Number analyzed (Participants) | 25 | 25
units on a scale, each item scored 0-4
  Pre Training Assessment | 44 (6) | 44 (4)
  Mid Training Assessment | 46 (6) | 46 (4)
  Post Training Assessment | 48 (4) | 48 (3)
  3 Month Post Training Assessment | 48 (4) | 48 (3)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed, before and after every data collection session, through study completion.
Arm/Group | Stride Management Assist (SMA) System | Impairment Based Therapy
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Intervention was limited to 6-8 weeks with a follow-up of 3 months. Determining if effects lasted more than 3 months and length of therapy needed to achieve long lasting effects is beneficial. A custom fitting SMA may enhance outcomes in users.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT01994395/Prot_SAP_000.pdf